CLINICAL TRIAL: NCT06924164
Title: Snappy Hip Trial: A Randomized Crossover Trial Comparing the Clinical and Cost-effectiveness of Progressive Resistance Training Compared to Usual Care on Pain for Adults With External Snapping Hip
Brief Title: Progressive Resistance Training for Adults With External Snapping Hip
Acronym: Snappy Hip
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Snappy Hip Tirial; 4308-00012B (Other Grant/Funding Number: Independent Research Fund Denmark)
Record Dates: First submitted 2025-03-28; First posted 2025-04-11 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: External Snapping Hip; Coxa Saltans External
Keywords: External snapping hip; Progressive resistance training; Coxa saltans external; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise Therapy; Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group: Wait and see approach (Other): The control group are randomized to 12 weeks of waiting time followed by 12 weeks of progressive resistance training.
  Interventions: Other: Progressive resistance training; Behavioral: Waiting time
- Intervention group: progressive resistance training (Experimental): The intervention group are randomized to 12 weeks of progressive resistance training followed by 12 weeks of self guided exercise
  Interventions: Other: Progressive resistance training; Behavioral: Self guided exercise

INTERVENTIONS:
Other: Progressive resistance training — The progressive resistance program consist of a five-minute aerobic warm-up on either an ergometer bike, treadmill or rowing machine followed by six resistance training exercises: landmine twist, walking lunges, leg press, hip abduction, hip adduction and hip flexion. All training sessions (three per week) will be supervised for the first two weeks. After that, there will be one weekly supervised training session and two self-directed sessions. The subjects will be scheduled for 36 training sessions over 12 weeks, of which 16 will be supervised. Each training session is designed based on the findings from the feasibility study and is expected to last approximately one hour. If a subject cannot perform all scheduled sessions in a week, additional sessions will be planned for the following week to obtain the 16 supervised sessions.
  Other Names: Exercise therapy
Behavioral: Waiting time — 12 weeks of waiting time
  Other Names: Waitlist; Wait
  Arms: Control group: Wait and see approach
Behavioral: Self guided exercise — 12 weeks of self guided exercise
  Other Names: Wait; Self training
  Arms: Intervention group: progressive resistance training

SUMMARY:
External snapping hip is characterised by an audible and painful snap during hip movement among physical active people around 15-40 years old. Progressive resistance training has been suggested as a new potential treatment path in treating patients with external snapping hip. The investigators conducted a feasibility study and found that patients reported less pain and improved their physical function, quality of life and muscle strength after 12 weeks of progressive resistance training. The overall aim of the project is to compare hip pain in patients with external snapping hip treated with progressive resistance training to a wait-and-see approach, in a randomised controlled trial. This study has the potential to establish a new and specific treatment option for patients with external snapping hip, to be used nationally and internationally.

DETAILED DESCRIPTION:
This trial is an international multicentre randomised controlled assessor-blinded crossover trial, following the CONSORT guidelines. The intervention is a 12-week progressive resistance training programme, and the trial is designed with three follow-up time points. After the baseline test, the patients will be randomised in a 1:1 ratio to either the intervention or the control group using the Research Electronic Data Capture (REDCap) source hosted at Aarhus University. For both groups, the first test will be the baseline test, conducted before the randomisation. The second test will be conducted 6 weeks after randomisation, the third test will be conducted 12 weeks after randomisation and the fourth and last test will be conducted 24 weeks after randomisation. The primary outcome will be the change from baseline to the third follow-up, and the trial will be powered based on this period. The lasting effect of the intervention will be evaluated from baseline to the fourth follow-up test for the intervention group.

ELIGIBILITY:
Inclusion criteria:

* Age 18-40 years (10)
* Experienced lateral hip joint "snapping" with pain discomfort within the last 14 days
* Able to demonstrate the audible and/or visible lateral "snapping" during lateral hip joint movementor popping sound when the hip joint moves
* Capable of commuting to the training facility
* Proficient in reading and understanding Danish or English

Exclusion criteria:

* Previous surgery on the affected hip
* Planned surgery on lower extremities within the trial period
* Anterior or medial hip discomfort that substantially exceeds the lateral hip discomfort
* Any contraindication to exercise
* Neurological, rheumatoid, or mental conditions affecting the hip function
* Ongoing active cancer treatment
* Planned vacation for more than 14 days within the intervention period
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
HAGOS Pain | Baseline, week 6, week 12 and week 24
  The HAGOS is a patient-reported questionnaire consisting of six different subscales. The pain subscale consists of 10 questions, which are all answered using standardised answer options following a 0-4-point Likert Scale. The scores are transformed into a subscale score ranging from 0 (worst) to 100 (best). A minimal clinically relevant difference of the HAGOS pain subscale has been reported to be 9.7 points among a group of patients undergoing hip arthroscopy for femoroacetabular impingement.

SECONDARY OUTCOMES:
HAGOS | Baseline, week 6, week 12 and week 24
  The remaining five subscales of HAGOS: symptoms, function in daily living (ADL), function in sport and recreation (Sports/Rec), participation in physical activities (PA) and hip and/or groin-related quality of life (QOL). The scores are transformed into a subscale score ranging from 0 (worst) to 100 (best).
UCLA-AS | Baseline, week 12 and week 24
  The patient-reported questionnaire: the University of California Los Angeles Activity Scale. There is only one question with 10 answers, ranging from 1 (worst) to 10 (best).
GPE | Baseline, week 12 and week 24
  The patient-reported questionnaire: the Global Perceived Effect, where the participant answers four questions about the effect of the treatment received. Each question has 7 possible answers, ranging from 1 (best) to 7 (worst).
Single leg hop test | Baseline, week 12 and week 24
  The objective measures include the single-leg hop for a distance test to test hip function. The hop distance is measured in cm.
30 second unilateral sit-to-stand test | Baseline, week 12 and week 24
  The unilateral 30 second Sit to Stand test (unilateral 30STS) is a clinical test of lower extremity function. The unilateral 30STS tests how many correct repetitions of a sit to stand from a chair, a participant can complete in 30 seconds.
Number of training sessions the participant participated in | Throughout the study, summed in week 24
  Adherence to the exercise protocol will be evaluated based on information from the physiotherapists and a self-reported training diary. Good adherence will be defined as participation in more than ≥70% of all training sessions (both supervised and self-training).
Adverse events | Throughout the study, summed in week 24
  The physiotherapist will record any adverse events occurring during the study period.

OTHER OUTCOMES:
EQ-5D-5L | Baseline, week 12 and week 24
  The patient-reported questionnaire: the European Quality of life 5 Dimensions with 5 Levels (EQ-5D-5L) where the participant answers six questions in relation to health-related quality of life
iPCQ | Baseline, week 12 and week 24
  The patient-reported questionnaire: the Productivity Costs Questionnaire, where information on productivity is collected .
HUQ | Baseline, week 12 and week 24
  Health Utilisation Questionnaire (HUQ) where information on healthcare and medicine is collected.
Usage of analgesics due to hip-related pain | Baseline, week 12 and week 24
  The participants will be asked if they take any analgesics due to hip-related pain. If yes, they will be further asked what type of medicine (Paracetamol/NSAID/Morfin/Other) and how often (Never/Monthly/Weekly/Daily).

CONTACTS AND LOCATIONS:
Overall Officials: Stig S Jakobsen, PhD, Study Director — Department of Orthopedic Surgery, Aarhus University Hospital, DK; Lisa U Tønning, MHSc, Principal Investigator — Department of Orthopedic Surgery, Aarhus University Hospital, DK; Inger Mechlenburg, DMSc, Study Director — Department of Clinical Medicine, Aarhus University, DK; Ulrik Dalgas, PhD, Study Director — Department of Public Health, Sports, Aarhus University, DK; Troels Kjeldsen, PhD, Study Director — Department of Orthopedic Surgery, Aarhus University Hospital, DK; Cara Lewis, PhD, Study Director — Department of Physical Therapy, Boston University, Boston, US; Martin Lamm, MSc, Study Director — Department of Orthopedic Surgery, Aarhus University Hospital, DK; Joanne L Kemp, PhD, Study Director — La Trobe Sport and Exercise Medicine Research Centre, La Trobe University, Melbourne, Australia
Locations (13):
- Denmark (13):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen
  - Bispebjerg og Frederiksberg Hospital, Copenhagen
  - Regionshospitalet Gødstrup, Herning
  - Nordsjællands Hospital - Hillerød, Hillerød
  - Regionshospitalet Horsens, Horsens
  - Hvidovre Hospital, Hvidovre
  - Sjællands Universitetshospital - Køge, Køge
  - Næstved, Slagelse og Ringsted Hospital, Næstved
  - Odense Universitetshospital, Odense
  - Regionshospitalet Randers, Randers
  - Sygehus Lillebælt - Vejle, Vejle

IPD SHARING:
Plan to Share IPD: Yes
Anonymized patient-level data will be made available if required by the scientific journal, in which the results of the trial are published. Additionally, researchers presenting a justified cause for receiving the data can obtain it after a data access agreement has been signed.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after publication of the trial upon reasonably request.
Access Criteria: Applications for data access will be reviewed by the author group. The applicant will be required to sign a data access agreement.